CLINICAL TRIAL: NCT02588313
Title: Investigation of Long-term Effects of CarelessTM on Microcirculation in Healthy Volunteers - a Randomized, Double-blind, Placebo-controlled Study With Parallel Design
Brief Title: Investigation of Long-term Effects of CarelessTM on Microcirculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital Solutions Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTS910/15
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2015-10

CONDITIONS: Disorder of Circulatory System; Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mango fruit powder 100mg (Active Comparator): Mango fruit powder 100mg
  Interventions: Dietary Supplement: Mango fruit powder
- Mango fruit powder 300mg (Active Comparator): Mango fruit powder 300mg
  Interventions: Dietary Supplement: Mango fruit powder
- Placebo formulation (Placebo Comparator): Placebo formulation
  Interventions: Dietary Supplement: Mango fruit powder

INTERVENTIONS:
Dietary Supplement: Mango fruit powder — Investigation of long-term effects of CarelessTM on microcirculation in healthy volunteers - a randomized, double-blind, placebo-controlled study with parallel design
  Other Names: CarelessTM

SUMMARY:
Aim of the study is to investigate long-term effects of CarelessTM, a Mangifera indica fruit powder on microcirculation and endothelial function after supplementation of 4 weeks. Effects will be investigated with 100mg and 300mg CarelessTM and compared to placebo.

DETAILED DESCRIPTION:
Aim of the study is to investigate long-term effects of CarelessTM, a Mangifera indica fruit powder on microcirculation and endothelial function after supplementation of 4 weeks. Effects will be investigated with 100mg and 300mg CarelessTM and compared to placebo.

To describe targeted parameter, cutaneous microcirculation will be measured at 1 mm depth as well as flow mediated endothelial function at the beginning and end of supplementation, each. Furthermore, the parameters will be determined postprandially 1 hour after glucose loading. Additionally the influence on the glucose metabolism, as well as on body weight and body fat will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Men and postmenopausal women
* HOMA Index ≥2 and <5
* BMI: 19 - 30 kg/m2
* Age ≥ 40 and ≤ 70 years
* Nonsmoker
* Written consent to participate in the study
* Able and willing to follow the study protocol procedures

Exclusion Criteria:

* Relevant history, presence of any medical disorder or chronic intake of medication/dietary sup-plements (e.g. polyphenols, L-Arginine, Niacin, medication of haemodilution, blood flow stimu-lating products like Aspirin (Acetylsalicylsäure), Clopidogrel (Adenosin-Diphosphat(ADP)-Inhibitors), Glykoprotein-IIb/IIIa-Inhibitors, Heparin, Marcumar (Vitamin K antagonists); Dabiga-tran (Faktor IIa synthese Inhibitors) Rivaroxaban (Faktor Xa Antagonist), Statins) potentially in-terfering with this study at screening.
* For this study clinically relevant abnormal laboratory, vital signs or physical findings at screening
* Diabetes
* Atopic dermatitis or affected skin at the forearm
* Injury on the finger, influencing the EndoPATTM measurement
* Regular consumption of caffeine > 275 mg (equivalent to 3-4 cups of coffee or 9 cups of black tea)
* Change of dietary habits within the 2 weeks prior to screening (for instance start of a diet high in vegetables and fruits (≥ 5 portions per day))
* Diet high in vegetables and fruits ≥ 5 portions per day
* Participants anticipating a change in their lifestyle or physical activity levels during the study.
* Subjects not willing to avoid polyphenol rich foods and abstain from beverages containing caf-feine the day prior to visit 1 and 2.
* Subjects not willing to abstain from intake of analgesic medication (e.g. Aspirin) 24 hours prior to and during visit 1 and 2.
* Sunbathing or the use of sun-beds 2 weeks prior to study days
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study.
* Known hypersensitivity to the study preparation or to single ingredients
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding sub-ject.
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study.
* Subject involved in any clinical or food study within the preceding month

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Measurement of circulation | Baseline at day 1 and after 4 weeks supplementation
  Measurement of dermal microcirculation using "O2C, Lea Technik":
  * Relative peripheral blood flow (LDF)
  * Venous oxygen saturation (SO2 ven)
  * Relative amount of haemoglobin (rHb). Delta change of dermal microcirculation from baseline to end of supplementation is investigated. Addi-tionally, the delta change of dermal microcirculation from baseline to end of supplementation post-prandial is determined, which means the evaluation of postprandial effects on reactive hyperaemia index after glucose load.

SECONDARY OUTCOMES:
Measurement of glucose related biomarker | Baseline at day 1 and after 4 weeks supplementation
  Measurement of Biomarker HOMA-Index, HbA1c at baseline and end of supplementation under fasting conditions.
Questionnaire on fatigue and vigor | Baseline at day 1 and after 4 weeks supplementation
  Questionnaire on fatigue and vigor
Monitoring of adverse effects | During study execution over 4 weeks
  Reporting of adverse effects to evaluate tolerability
Measurement of endothelial function using "EndoPATTM, Itamar" | Baseline at day 1 and after 4 weeks supplementation
  Measurement of endothelial function using "EndoPATTM, Itamar"
  * Reactive hyperaemia index (RHI and lnRHI)
  * Arterial stiffness (AI75) Delta change of endothelial function and arterial stiffness from baseline to end of supplementation is investigated. Additionally, the delta change of endothelial function from baseline to end of supplemen-tation postprandial is determined, which means the evaluation of postprandial effects on relative hy-peraemia index after glucose load.
Measurement of ox LDL | Baseline at day 1 and after 4 weeks supplementation
  Measurement of ox LDL

OTHER OUTCOMES:
Body composition | Baseline at day 1 and after 4 weeks supplementation
  Body weight and body fat (Body impedance analysis) determination
Blood glucose | Baseline at day 1 and after 4 weeks supplementation, before 1h and 2h after glucose loading
  Capillary blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Reule, PhD, Study Chair — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany